CLINICAL TRIAL: NCT05143918
Title: Assessment of Quality of Life Among Hypothyroid Patients in Assiut University Hospitals
Brief Title: Quality of Life Among Egyptian Hypothyroid Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Fathy Radwan Abd El Zaher, Physician at internal medicine department at Assiut University Hospital, Assiut University
Other Study IDs: quality of life
Record Dates: First submitted 2021-11-23; First posted 2021-12-03 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism, Egypt, Quality of life
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypothyroid patients as a cases: 1. Inclusion criteria:
     1. age ranges will be 18 - 60 years
     2. both genders
     3. previously confirmed diagnosed
  2. Exclusion criteria:
     1. pregnancy
     2. other comorbidities (hypertension, diabetes, malignancy,,,etc)
  Interventions: Other: assessment of quality of life using questionnaire
- Control group: Healthy people without chronic disease
  Interventions: Other: assessment of quality of life using questionnaire

INTERVENTIONS:
Other: assessment of quality of life using questionnaire — assessment of quality of life in hypothyroid patients using SF 36 questionnaire

SUMMARY:
Assessment of quality of life among hypothyroid patients in Assiut University Hospital

DETAILED DESCRIPTION:
Hypothyroidism is an underactive thyroid gland. Hypothyroidism means that the thyroid gland can't make enough thyroid hormone to keep the body running normally. People are hypothyroid if they have too little thyroid hormone in the blood. Common causes are Iodine deficiency, autoimmune disease, such as Hashimoto's thyroiditis, surgical removal of the thyroid, and radiation treatment.

There are three types of hypothyroidism: primary, secondary and tertiary. Primary hypothyroidism results from a low level of thyroid hormone due to destruction of the thyroid gland. This condition results in increased secretion and elevation of serum thyroid-stimulating hormone (TSH) levels. If the structure of the gland remains normal, dysfunction can be caused by decreased TSH secretion from the pituitary; this Is called secondary hypothyroidism.

In tertiary hypothyroidism, a decrease in thyroid hormone arises from inadequate secretion of thyrotropin-releasing hormone (TRH) from the hypothalamus. It is not always possible to differentiate between secondary and tertiary hypothyroidism, and they are often collectively referred to as central hypothyroidism. About 99%ofhypothyroidism cases are primary hypothyroidism.

Hypothyroidism is common throughout the world. In iodine-sufficient countries, the prevalence of hypothyroidism ranges from 1% to 2%. rising to 7% in individuals aged between 85 and 89 years. In the absence of age-specific reference ranges for TSH, an ageing population is likely to result in a higher prevalence of hypothyroidism. Hypothyroidism is approximately ten times more prevalent in women than men10. the awareness of hypothyroidism has increased gradually, as has rate of initiation of levothyroxine substitution.

Symptoms usually develop slowly and the patient may not realise to have a medical problem for several years. Common symptoms include: tiredness, being sensitive to cold, weight gain, constipation, depression, slow movements and thoughts, muscle aches and weakness, muscle cramps, dry and scaly skin, brittle hair and nails, loss of libido (sex drive), pain, numbness and a tingling sensation in the hand and fingers (carpal tunnel syndrome),irregular periods or heavy periods.

Health-related quality of life (HRQL) is a subjective assessment of the effects of disease and its treatment on the physical, social, psychological, and somatic dimensions of a patient's life. Thus, HRQL is considered an important supplementary outcome measure in the management of different conditions.

Thyroid hormones are important for the body's total energy metabolism and the neuroendocrine function. Hence, it seems apparent that a dysfunction of the thyroid hormone secretion should have a major influence on the total capacity of the body, both physically and mentally. Increasing attention is being paid to assessing HRQL among patients with thyroid disorders, and previous studies have revealed that HRQL is frequently affected in patients with hypothyroidism.

Up to our knowledge, no previous study explored the quality of life and its correlates among Egyptian hypothyroidism patients. The current study aims to assess the quality of life and its predictor among hypothyroidism in Assiut University Hospital

ELIGIBILITY:
Inclusion Criteria:

1. age ranges will be 18 - 60 years
2. both genders
3. previously confirmed diagnosed

Exclusion Criteria:

* Exclusion criteria:

  1. pregnancy
  2. other comorbidities (hypertension, diabetes, malignancy,,,etc)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cases as hypothyroid patients and healthy control
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
predictors of quality of life among hypothyroid patients | nearly two year
  Using the Short Form (36) Health Survey (SF-36) questionnaire all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100.

CONTACTS AND LOCATIONS:
Overall Officials: Nabawia M Tawfik, Study Chair — Assiut University; Ghada Abd El Rahman, Study Director — Assiut University; Doaa M Osman, Study Director — Assiut University; Noha F Radwan, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shivaprasad C, Rakesh B, Anish K, Annie P, Amit G, Dwarakanath CS. Impairment of Health-related Quality of Life among Indian Patients with Hypothyroidism. Indian J Endocrinol Metab. 2018 May-Jun;22(3):335-338. doi: 10.4103/ijem.IJEM_702_17. PMID 30090724
- [Background] Blazewicz A, Wisniewska P, Skorzynska-Dziduszko K. Selected Essential and Toxic Chemical Elements in Hypothyroidism-A Literature Review (2001-2021). Int J Mol Sci. 2021 Sep 20;22(18):10147. doi: 10.3390/ijms221810147. PMID 34576309
- [Background] Taylor PN, Albrecht D, Scholz A, Gutierrez-Buey G, Lazarus JH, Dayan CM, Okosieme OE. Global epidemiology of hyperthyroidism and hypothyroidism. Nat Rev Endocrinol. 2018 May;14(5):301-316. doi: 10.1038/nrendo.2018.18. Epub 2018 Mar 23. PMID 29569622
- [Result] Mitchell AL, Hegedus L, Zarkovic M, Hickey JL, Perros P. Patient satisfaction and quality of life in hypothyroidism: An online survey by the british thyroid foundation. Clin Endocrinol (Oxf). 2021 Mar;94(3):513-520. doi: 10.1111/cen.14340. Epub 2020 Dec 17. PMID 32978985
- See also: Related Info — http://www.nhs.uk/conditions/underactive-thyroid-hypothyroidism/symptoms/